CLINICAL TRIAL: NCT03294980
Title: Chronic Lymphoid Leukaemia Observatory in Finistere Area, France
Acronym: OFICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: OFICE
Record Dates: First submitted 2016-08-26; First posted 2017-09-27 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Chronic Lymphoid Leukaemia
Keywords: Chronic lymphocytic leukemia; Observational study
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cell pellet More than 95% CD5+CD19+ lymphocytes

SUMMARY:
Brief Summary: The purpose of the OFICE registry is to characterize and describe the CLL patients' population from the Finistere area and evaluates the association between different patient characteristics, prognosis and treatment patterns.

Detailed Description: OFICE is a single center, prospective, observational registry of CLL patients designed to provide a general description of the CLL patients' population from the Finistere area, France. The registry will also provide information on the association of cytogenetic and immunophenotypic characteristics with disease progression, as well as treatment patterns and healthcare resource utilization. These data will be accessible and beneficial for researchers and physicians and will help guide clinical practice and future clinical or fundamental studies.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Clinical diagnosis of CLL/SLL that meets published diagnostic criteria (Hallek 2008)
* Willing and able to provide informed consent
* Willing and able to provide blood sample at time of enrollment

Exclusion Criteria:

* Diagnosis of other B-cell malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Chronic Lymphoid Leukaemia
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-11; Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence | Year 0 (Y)
  Clinical data

SECONDARY OUTCOMES:
Incidence | Year 0
  Clinical and biological data
Description of baseline clinical-biological | Year 0, Year 1, Year 2, Year 3
  Clinical data, complete blood count, Matutes score and parameters, cytogenetic, IgVH mutations, CD38 (%), medical treatment will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Yves Reanudineau, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Derived] Marlin A, Le Pape F, Troadec T, Le Goff J, Tripier R, Berthou C, Patinec V. Zn2+ triazamacrocyclic chelators with methylpyridine pendant arms for B-cell apoptosis: a structure-activity study. Dalton Trans. 2025 Feb 25;54(9):3939-3951. doi: 10.1039/d4dt02962c. PMID 39895421
- [Derived] Debant M, Burgos M, Hemon P, Buscaglia P, Fali T, Melayah S, Le Goux N, Vandier C, Potier-Cartereau M, Pers JO, Tempescul A, Berthou C, Bagacean C, Mignen O, Renaudineau Y. STIM1 at the plasma membrane as a new target in progressive chronic lymphocytic leukemia. J Immunother Cancer. 2019 Apr 23;7(1):111. doi: 10.1186/s40425-019-0591-3. PMID 31014395
- [Derived] Bagacean C, Tempescul A, Ternant D, Banet A, Douet-Guilbert N, Bordron A, Bendaoud B, Saad H, Zdrenghea M, Berthou C, Paintaud G, Renaudineau Y. 17p deletion strongly influences rituximab elimination in chronic lymphocytic leukemia. J Immunother Cancer. 2019 Jan 29;7(1):22. doi: 10.1186/s40425-019-0509-0. PMID 30696487